CLINICAL TRIAL: NCT04075539
Title: Home-based Cycling Using Connected Ergometric Bicycles for People With Lumbar Spinal Stenosis: a Randomized Controlled Trial
Brief Title: Home-based Cycling for People With Lumbar Spinal Stenosis
Acronym: FLEXCAL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P160147; 2023-A00601-44 (Other: ID-RCB)
Record Dates: First submitted 2019-08-29; First posted 2019-08-30 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Symptomatic Lumbar Spinal Stenosis
Keywords: Lumbar spinal stenosis; Neurogenic claudication; Low back pain; Exercise therapy; Endurance training; Cycling; Randomized trial
MeSH Terms: conditions — Spinal Stenosis; Low Back Pain

STUDY DESIGN:
Masking Description: single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based cycling program associated to usual care (Experimental)
  Interventions: Other: Home-based cycling program
- Outpatient physiotherapy (Other)
  Interventions: Other: usual care

INTERVENTIONS:
Other: Home-based cycling program — Usual care (i.e. standardized prescription of 6 sessions of outpatient physiotherapy), and
  * 1 supervised session of cycling aimed at explaining how to use the connected ergometric bicycle and at designing a personalized home-based cycling program
  * a 12-month home-based cycling program using connected ergometric bicycles which intensity and dose are self-determined
  * 3 phone or email contacts with a care provider to deliver positive feedbacks and encouragements
  Arms: Home-based cycling program associated to usual care
Other: usual care — A prescription of 6 sessions of outpatient physiotherapy
  Arms: Outpatient physiotherapy

SUMMARY:
The main objective of the study is to compare the efficacy on back-specific activity limitations at 4 months after-randomisation of home-based cycling using connected ergometric bicycles associated with usual care to usual care.

DETAILED DESCRIPTION:
Lumbar spinal stenosis is a prevalent and disabling condition in elderly people. Lumbar spinal stenosis results in back and leg pain when standing and walking (radicular claudication), while symptoms regress in sitting position. The inability to stand or walk significantly impairs functioning and health-related quality of life of elders, and has an important healthcare cost.

The 2 main treatment options for lumbar spinal stenosis are conservative or surgical treatments. Previous data suggested that laminectomy may be more effective on pain and function than conservative therapy. However, the benefit-risk balance of surgery should be carefully considered in this population with numerous co-morbidities, and evidence is inconsistent. Therefore, conservative therapy is usually the first line option. Data regarding exercise therapy are scarce. Flexion-based exercises are usually recommended. A pilot study suggested that flexion-based endurance training program, namely cycling, could be an effective and safe method to improve pain, function and health-related quality of life in elderly people with chronic lumbar pain. However, barriers to adhering to the program were detected and might have influenced clinical endpoints. Non-pharmacological interventions in spinal conditions are not 'one-size-fits-all' and measures to enhance adherence have to be applied.

The hypothesis is that home-based cycling using connected ergometric bicycles associated with usual care could be more effective than usual care in reducing back-specific activity limitations at 4 months in people with lumbar spinal stenosis.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 50 year-old
* radicular claudication (i.e. walking-induced low back, buttock and/or leg pain, relieved in siting and/or lumbar flexion positions) diagnosed by a physician
* MRI or CT-scan findings consistent with LSS reported on a written radiology report provided by a board-certified radiologist or a resident in radiology

Exclusion Criteria:

* inability to speak and/or read French language
* inability or refusal to perform ergometric bicycle at home
* patients already having an ergometric bicycle at home
* history of lumbar spine surgery in the previous 12 months
* cognitive disorders
* severe neurologic or vascular disorders involving the lower limbs
* contraindication to a rehabilitation program assessed by medical examination
* people under tutorship or curatorship
* protected adults

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Change in back-specific activity limitations | 4 months after-randomization
  Mean change from baseline in mean back-specific activity limitations in the previous month using the self-administered Oswestry Disability Index (ODI) total score (0 no limitations and 100 maximal limitations).

SECONDARY OUTCOMES:
Change in maximal walking distance | 4 months post-randomization
  Mean change from baseline in mean maximal walking distance (meters) using an adapted version of the self-paced walking-test
Change in lumbar pain | 4, 6 and 12 months post-randomization
  Mean change from baseline in mean low back pain intensity in the previous 48 hrs on a self-administered 11-point pain numeric rating scale (0 no pain and 100 maximal pain)
Change in radicular pain | 4, 6 and 12 months post-randomization
  Mean change from baseline in mean radicular pain intensity in the previous 48 hrs on a self-administered 11-point pain numeric rating scale (0 no pain and 100 maximal pain)
Change in the physical component of health-related quality of life | 4, 6 and 12 months post-randomization
  Mean change from baseline in the mean physical component of health-related quality of life assessed by the physical component score of the self-administered 12-Item Short Form Survey (9.95 worst possible and 70.02 best possible)
Change in lumbar spinal stenosis-specific activity limitations | 4, 6 and 12 months post-randomization
  Mean change from baseline in mean LSS-specific activity limitations using the physical function subscore of the self-administered Zurich Claudication Questionnaire (1 no limitations and 4 maximal limitations)
Change in back-specific activity limitations | 6 and 12 months post-randomization
  Mean change from baseline in mean spine-specific activity limitations assessed by the total score of the self-administered Oswestry Disability Index (0 no limitations and 100 maximal limitations)
Percentage of patients who undergo spinal surgery | From baseline to 12 months post-randomization
  Self-reported spinal surgery for lumbar spinal stenosis

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Nguyen, MD, PhD, Principal Investigator — Université de Paris, Faculté de Médecine Paris Descartes; François Rannou, MD, PhD, Study Director — Université de Paris, Faculté de Médecine Paris Descartes; Isabelle Boutron, MD, PhD, Study Chair — Université de Paris, Faculté de Médecine Paris Descartes
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Service de Rééducation et de Réadaptation de l'Appareil Locomoteur et des Pathologies du Rachis, Hôpital Cochin, Paris, Île-de-France Region, France

REFERENCES:
- [Background] Nguyen C, Boutron I, Roren A, Baron G, Pauwels C, Lefevre-Colau MM, Poiraudeau S, Dupeyron A, Coudeyre E, Rannou F. Home-based cycling using connected ergometric bicycles for people with lumbar spinal stenosis (FLEXCAL): Protocol for a randomised trial. Ann Phys Rehabil Med. 2021 Mar;64(2):101351. doi: 10.1016/j.rehab.2019.12.006. Epub 2020 Jan 23. No abstract available. PMID 31982599